CLINICAL TRIAL: NCT03697993
Title: Multi-center, Randomized, Open-label Trial to Evaluate the Efficacy of Oral Fosfomycin Versus Oral Levofloxacin Strategies in Complicated Urinary Tract Infections (FOCUS)
Brief Title: Safety and Efficacy Study of Oral Fosfomycin Versus Oral Levofloxacin to Treat Complicated Urinary Syndromes (FOCUS)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate enrollment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0045; HHSN272201300018I
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2018-09-11

CONDITIONS: Urinary Tract Infection
Keywords: Fosfomycin; levofloxacin; Open-label; Phase IV; UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin; Levofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strategy 1 (Experimental): Fosfomycin 3 g orally once daily for 5-7 days as initial or step-down oral therapy for complicated urinary tract infections (cUTI) without bacteremia with a uropathogen after 0-48 hours of parenteral antibiotic therapy, and if indicated a subsequent investigator-directed adjustment to another adequate oral therapy. N=317
  Interventions: Drug: Fosfomycin tromethamine
- Strategy 2 (Experimental): Levofloxacin 750 mg orally once daily for 5-7 days as initial or step-down oral therapy for cUTI without bacteremia with a uropathogen after 0-48 hours of parenteral antibiotic therap, and if indicated a subsequent investigator-directed adjustment to another adequate oral therapy.y. N=317
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Fosfomycin tromethamine — Administered orally as 3-gram single-dose sachet into 3-4 ounces (1 / 2 cup) of cool water; each dose must be taken immediately after dissolving in water. Hot water should not be used to dissolve fosfomycin. It may be taken either with or without food for normal kidney function. If Creatinine Clearance (CrCl) is less than 20 mL/min, fosfomycin should be taken as 3 grams every other day.
  Arms: Strategy 1
Drug: Levofloxacin — 750 mg is administered orally as one tablet once daily with or without food for normal kidney function. If Creatinine Clearance (CrCl) is 20-49 mL/min, 750 mg should be taken every other day. If on subsequent testing post-randomization, the Creatinine Clearance (CrCl) is less than 20 mL/min, followed by the dose is 500 mg every other day.
  Arms: Strategy 2

SUMMARY:
This is a Phase 4, multi-center, open-label, randomized pragmatic superiority clinical trial comparing two strategies for initial or step-down oral therapy for complicated urinary tract infections (cUTI) after 0-48 hours of parenteral antibiotic therapy. The trial will evaluate the success and safety of a strategy of initial or step-down fosfomycin, administered at a dose of 3 g once daily, vs. a strategy of initial or step-down levofloxacin administered at a dose of 750 mg once daily. Investigator-directed adjustment to another adequate oral therapy is allowed 1) if the causative pathogen is not susceptible in vitro to quinolone initial or step-down therapy in a subject randomized to the levofloxacin strategy, OR 2) if the subject develops an intolerance or allergy to the initial step-down oral therapy and at the investigator's discretion, OR 3) the subject has an underlying condition posing increasing risk for adverse events from quinolone therapy. The duration of oral therapy (initial + investigator-directed adjustment if indicated) in each strategy is 5-7 days of any per protocol antibiotic to which the pathogen is susceptible. The dosing of oral therapy depends on creatinine clearance (CrCl). The trial will enroll approximately 634 patients that are either male or female aged 18 or older with cUTI from outpatient and inpatient settings. The study will take place over 25 months in up to 15 US sites. The primary objective is to compare Strategy 1 and Strategy 2 in terms of treatment success rates at Test of Cure (TOC).

DETAILED DESCRIPTION:
This is a Phase 4, multi-center, open-label, randomized pragmatic superiority clinical trial comparing two strategies for initial or step-down oral therapy for complicated urinary tract infections (cUTI) without bacteremia with a uropathogen after 0-48 hours of parenteral antibiotic therapy. The trial will evaluate the success and safety of a strategy of initial or step-down fosfomycin, administered at a dose of 3 g once daily, vs. a strategy of initial or step-down levofloxacin administered at a dose of 750 mg once daily. Investigator-directed adjustment to another adequate oral therapy is allowed 1) if the causative pathogen is not susceptible in vitro to quinolone initial or step-down therapy in a subject randomized to the levofloxacin strategy, OR 2) if the subject develops an intolerance or allergy to the initial step-down oral therapy and at the investigator's discretion, OR 3) the subject has an underlying condition posing increasing risk for adverse events from quinolone therapy. The duration of oral therapy (initial + subsequent if indicated) in each strategy is 5-7 days of any per protocol antibiotic to which the pathogen is susceptible. The dosing of oral therapy depends on creatinine clearance (CrCl). The trial will enroll approximately 634 patients that are either male or female aged 18 or older with cUTI from outpatient and inpatient settings. The study will take place over 25 months in up to 15 US sites. The primary objective is to compare Strategy 1 and Strategy 2 in terms of treatment success rates at Test of Cure (TOC). The secondary objectives are: 1) to assess the safety of Fosfomycin; 2) to compare Strategy 1 and Strategy 2 in terms of solicited adverse events; 3) to compare Strategy 1 and Strategy 2 in terms of treatment success rates at End of Therapy (EOT).

ELIGIBILITY:
Inclusion Criteria:

1. Have documented clinical signs and/or symptoms of complicated urinary tract infection (cUTI) at diagnosis*.

   *Clinical signs and symptoms of cUTI include either:
   1. Pyelonephritis, as indicated by at least 2 of the following:

      * Documented fever (temperature greater than 38 degrees Celsius) accompanied by symptoms of rigors, chills, or "warmth"
      * Flank pain
      * Costovertebral angle tenderness on physical exam
      * Nausea or vomiting
      * Dysuria, urinary frequency, or urinary urgency OR
   2. Complicated lower UTI, as indicated by at least 2 of the following new or worsening symptoms of cUTI:

      * Dysuria, urinary frequency, or urinary urgency
      * Documented fever (temperature greater than 38 degrees Celsius) accompanied by symptoms of rigors, chills, or "warmth"
      * Documented hypothermia (temperature less than 35.5 degrees Celsius)
      * Suprapubic pain or pelvic pain
      * Suprapubic tenderness on physical exam
      * New onset of foul smell to urine or increased cloudiness of urine per subject or their caregiver
      * Nausea or vomiting

   AND at least 1 of the following complicating factors:
   * Males with documented history of urinary retention
   * Indwelling urinary catheter that is planned to be removed or replaced during study therapy and before End of Therapy (EOT)
   * Current obstructive uropathy that is scheduled to be medically or surgically relieved during study therapy and before End of Therapy (EOT)
   * Any functional or anatomical abnormality of the urogenital tract (including anatomic malformations or neurogenic bladder) with voiding disturbance resulting in at least 100 mL of residual urine OR with the need for intermittent or ongoing self-catheterization.
2. Able to understand and provide written informed consent*. *A legally acceptable representative may provide consent if the subject is unable to do so, provided this is approved by local institution-specific guidelines.
3. Anticipated to be able to be stepped down or initially started on study oral antibiotic therapy within 48 hours of enrollment*,**.

   *The readiness of a subject for initial or step-down oral therapy is determined by the primary medical team. In addition, for step down therapy the following conditions have to be met: temperature at randomization must be less than 38 degrees Celsius without any rigors/chills AND the subject must have an improvement in baseline symptoms of cUTI and no new cUTI symptoms.

   **Subject may be enrolled if he/she received a non-study oral antibiotic only if it is followed by parenteral antibiotics for less than 48 hours prior to de-escalation with study drugs.
4. Male or non-pregnant female.
5. Aged 18 years or older.
6. Women of childbearing potential* must agree to use an effective method of contraception** for the duration of the trial.

   *Female is considered of childbearing potential unless postmenopausal, or surgically/non surgically sterilized and at least 3 months has passed since sterilization procedure. A woman is considered postmenopausal if her last menstrual period was greater than or equal to 12 months.

   **Includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for greater than or equal to 180 days before the subject receiving the first dose of study drug, barrier methods such as condoms or diaphragms, effective intrauterine devices, NuvaRing (R), and licensed hormonal methods such as implants, injectables but not oral contraceptives.
7. If female of childbearing potential*, a negative urine or serum pregnancy test within 48 hours of randomization.

   *Female is considered of childbearing potential unless postmenopausal, or surgically/non surgically sterilized and at least 3 months has passed since sterilization procedure. A woman is considered postmenopausal if her last menstrual period was greater than or equal to 12 months.
8. Have pyuria (WBC count greater than or equal to 10/µL in unspun urine or greater than or equal to 10 per high power field in spun urine) or dipstick analysis positive (excluding "trace") for leukocyte esterase.
9. Have a pretreatment baseline urine culture specimen obtained within 48 hours before the first dose of any antibiotic is administered (including pre-study antibiotics)*.

   *Subjects may be enrolled in the trial and start study drug before the investigator knows the results of the baseline urine culture.
10. Able to reliably take, tolerate, and absorb oral medications, at the investigator's discretion.
11. Ability to understand study procedures and willing and able to comply with all required procedures and visits for the duration of the trial.

Exclusion Criteria:

1. Have a documented history of any moderate or severe hypersensitivity or allergic reaction to all five oral therapy options.
2. Have a concomitant infection at the time of randomization, which requires non-study systemic antibacterial therapy effective against complicated Urinary Tract Infection (cUTI) in addition to study drug.
3. Have received more than 48 hours of a potentially therapeutic antibiotic for treatment of the current cUTI within 72 hours before randomization*.

   *Except if the following apply:
   1. The subject has a known baseline urinary pathogen (urine culture positive) and has failed prior therapy clinically (persistence of inclusion criteria) AND
   2. The pathogen is known to be non-susceptible to the previous therapeutic regimen used or the urine culture remains positive with a density of greater than or equal to 50,000 CFU/mL or greater than or equal to 10,000 for catheterized patients.
4. Women breastfeeding or donating breast milk.
5. Have intractable UTI infection at baseline that the investigator anticipates would require more than 7 days of study drug therapy.
6. Have complete, permanent obstruction of the urinary tract*.

   *Patients with complete permanent obstruction expected to be medically or surgically treated prior to End of Treatment (EOT) are eligible.
7. Have confirmed fungal UTI at time of randomization (with greater than or equal to 10^3 fungal CFU/mL).
8. Have suspected or confirmed perinephric or intrarenal abscess.
9. Have suspected or confirmed prostatitis, epididymitis.
10. Have an ileal loop or known vesico-ureteral reflux.
11. Have a current urinary catheter that is not scheduled to be replaced before EOT*.

    *Intermittent straight catheterization or replacement of new nephrostomy catheters is acceptable.
12. Have planned inpatient urological intervention(s) for suspected infected kidney stone or any other planned urological procedure with anticipated antibiotic prophylaxis between randomization and End of Treatment (EOT).
13. Have bacteremia with a uropathogen causing cUTI.
14. Have an estimated or calculated Creatinine Clearance (CrCl) less than or equal to 20 mL/min or currently receiving hemo- or peritoneal dialysis at screening.
15. Have any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the subject or the quality of study data*.

    *Including any rapidly progressing disease or immediately life-threatening (acute hepatic failure, respiratory failure or septic shock).
16. Have participated in any interventional trial of an investigational product within 30 days before the proposed first day of study drug administration.
17. Plans to participate or currently enrolled in any interventional study of an investigational agent for the duration of the trial.
18. Previous randomization in this trial.
19. Any recent (less than 4 weeks) history of trauma to the pelvis or urinary tract.
20. Prior fosfomycin use in the past 12 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of California Los Angeles - Olive View Medical Center, Sylmar, California
  - Harbor UCLA Medical Center - Medicine - Infectious Diseases, Torrance, California
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Northwestern Medicine - Department of Obstetrics and Gynecology - Division of Female Pelvic Medicine and Reconstructive Surgery, Chicago, Illinois
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Infectious Disease Consultants - Wichita, Wichita, Kansas
  - Brigham and Women's Hospital - Infectious Diseases, Boston, Massachusetts
  - Henry Ford Health System - Henry Ford Hospital, Detroit, Michigan
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - U. of New Mexico Health Sciences Center - Dept. of Emergency Medicine, Albuquerque, New Mexico
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York
  - The Miriam Hospital - Infectious Diseases and Immunology Center, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were males and non-pregnant females aged >=18 years and diagnosed with complicated urinary tract infections (cUTIs) without bacteremia with a uropathogen. Participants were enrolled between 14NOV2018 and 03OCT2019.
Groups:
- Strategy 1: Fosfomycin 3 grams oral powder once daily for 5-7 days as initial or step-down oral therapy for cUTI without bacteremia with a uropathogen after 0-48 hours of parenteral antibiotic therapy, and if indicated a subsequent investigator-directed adjustment to another adequate oral therapy.
  Investigator-directed adjustment to another adequate oral therapy is allowed if the subject develops an intolerance or allergy to the initial step-down oral therapy and at the investigator's discretion, OR the subject has an underlying condition posing increased risk for adverse events from quinolone therapy. The duration of oral therapy (initial + subsequent if indicated) in each strategy is 5-7 days of any per protocol antibiotic to which the pathogen is susceptible. The dosing of oral therapy depends on creatinine clearance (CrCl).
  Another adequate oral therapy is defined as an oral therapy to which the pathogen shows in-vitro susceptibility AND to which the subject is tolerant based on history AND which is listed below:
  * Levofloxacin 750 mg oral tablet once daily (Strategy 1 only)
  * Amoxicillin-clavulanate 875/125 mg oral tablet twice daily
  * Cefixime 400 mg oral tablet once daily
  * Trimethoprim-sulfamethoxazole (TMP-SMX 160/800 mg) double-strength oral tablet twice daily
- Strategy 2: Levofloxacin 750 mg oral tablet once daily for 5-7 days as initial or step-down oral therapy for cUTI without bacteremia with a uropathogen after 0-48 hours of parenteral antibiotic therapy, and if indicated a subsequent investigator-directed adjustment to another adequate oral therapy.
  Investigator-directed adjustment to another adequate oral therapy is allowed if the causative pathogen is not susceptible in vitro to quinolone initial or step-down therapy in a subject randomized to the levofloxacin strategy, OR if the subject develops an intolerance or allergy to the initial step-down oral therapy and at the investigator's discretion. The duration of oral therapy (initial + subsequent if indicated) in each strategy is 5-7 days of any per protocol antibiotic to which the pathogen is susceptible. The dosing of oral therapy depends on creatinine clearance (CrCl).
  Another adequate oral therapy is defined as an oral therapy to which the pathogen shows in-vitro susceptibility AND to which the subject is tolerant based on history AND which is listed below:
  * Fosfomycin 3 grams oral powder once daily (Strategy 2 only)
  * Amoxicillin-clavulanate 875/125 mg oral tablet twice daily
  * Cefixime 400 mg oral tablet once daily
  * Trimethoprim-sulfamethoxazole (TMP-SMX 160/800 mg) double-strength oral tablet twice daily
Period: Overall Study
Arm/Group | Strategy 1 | Strategy 2
Started | 32 | 30
Initiated Treatment | 30 | 28
Switched Treatment (All participants who switched treatment within a strategy switched before initiation of the original treatment.) | 0 | 6 (Five (5) participants switched to Fosfomycin; 1 participant switched to Cefixime.)
Treated With at Least Two Dose of Fosfomycin | 27 | 4
Completed | 22 | 25
Not Completed | 10 | 5
Not completed — Became Ineligible after Enrollment | 1 | 3
Not completed — Enrolled but Treatment not Administered | 2 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Initial Urine Culture Negative | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Strategy 1 | Strategy 2 | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (19.4) | 46.3 (20.7) | 46.1 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 28 | 26 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 16 | 31
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62
cUTI [Count of Participants; unit: Participants]
  Pyelonephritis | 29 | 25 | 54
  Other cUTI | 3 | 5 | 8
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.02 (7.52) | 29.29 (8.65) | 28.12 (8.10)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Treatment Success at Test of Cure (TOC)
Description: Treatment success is defined as a combination of clinical cure and microbiological success.
  Clinical cure is defined as: 1) Resolution of UTI symptoms from presentation and 2) No new UTI symptoms and 3) Avoidance of parenteral antibiotic therapy, in or out of hospital, at any time after randomization OR oral antibiotic therapy different from per protocol.
  Microbiological success is defined as a reduction of the pathogen found at presentation to <10^4 CFU/mL for non-catheter specimens or <10^3 for catheter specimens on urine culture.
  A TOC visit was scheduled at 21 days (+7 days) after randomization.
Time Frame: Day 21
Population: The microbiologic Intention-to-Treat population includes all randomized participants who have a positive baseline bacterial culture of urine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 24 | 27
percentage of participants | 55 [36 to 73] | 73 [54 to 86]
Statistical Analysis 1: Comparison: Strategy 1 vs Strategy 2; Test type: Other; p = 0.264, Multiple imputation using Wald method; Risk Difference (RD) = -18, 95% CI 2-sided [-43.4 to 8.7]

2. Secondary Outcome: Number of Participants Reporting Solicited Adverse Events (AEs) Grade 2 and Above Among Those Who Received Fosfomycin
Description: Solicited AEs are AEs that are common following administration of these types of antibiotics. The solicited AEs were collected after first dose of study product was given and until the end of therapy (EOT). If subject is on fosfomycin, solicited AEs were collected for 2 days after last dose of fosfomycin or until EOT, whichever occurs last. The solicited AEs includes insomnia, headache, dizziness, nausea, vomiting, constipation, diarrhea, back pain, rhinitis, pharyngitis, allergic reaction, and candidiasis.
Time Frame: Day 1 through Day 12
Population: The fosfomycin safety population includes all subjects treated with at least two doses of fosfomycin.
Measure: Count of Participants; unit: Participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 27 | 4
Participants | 19 | 4

3. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs) Grade 2 and Above Among Those Who Received Fosfomycin
Description: The unsolicited AEs were collected in participants who received at least two doses of Fosfomycin from the time of second dose of Fosfomycin until the end of therapy (EOT) or 2 days after last dose of Fosfomycin, whichever occurs last.
Time Frame: Day 1 through Day 12
Population: The fosfomycin safety population includes all subjects treated with at least two doses of fosfomycin.
Measure: Count of Participants; unit: Participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 27 | 4
Participants | 2 | 0

4. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Among Those Who Received at Least Two Doses of Fosfomyci
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. Events are included if deemed by the investigator to be related to the study product. SAEs were only recorded in participants receiving at least two doses of fosfomyci.
Time Frame: Day 1 through Day 21
Population: The Fosfomycin safety population includes all subjects treated with at least two doses of Fosfomycin.
Measure: Count of Participants; unit: Participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 27 | 4
Participants | 2 | 0

5. Secondary Outcome: Percentage of Participants Reporting Solicited Adverse Events (AEs)
Description: as for outcome 2
Time Frame: Day 1 through Day 21
Population: The safety population includes all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 30 | 28
percentage of participants | 67 [48.8 to 80.8] | 68 [49.3 to 82.1]
Statistical Analysis 1: Comparison: Strategy 1 vs Strategy 2; Test type: Other; p = 1.000, Fisher Exact; Risk Difference (RD) = -1, 95% CI 2-sided [-26.2 to 24.3]

6. Secondary Outcome: Percentage of Participants Reporting Solicited Adverse Events (AEs) by Severity
Description: as for outcome 2
Time Frame: Day 1 through Day 21
Population: The safety population includes all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 30 | 28
percentage of participants
  Moderate | 53 [36 to 70] | 50 [33 to 67]
  Severe | 13 [5 to 30] | 18 [8 to 36]
Statistical Analysis 1: Comparison: Strategy 1 vs Strategy 2; Test type: Other; p = 0.894, Proportional odds model using Wald test; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 2.5]

7. Secondary Outcome: Percentage of Participants Achieving Treatment Success at End of Therapy (EOT)
Description: Treatment success is defined as a combination of clinical cure and microbiological success.
  Clinical cure is defined as: 1) Resolution of UTI symptoms from presentation and 2) No new UTI symptoms and 3) Avoidance of parenteral antibiotic therapy, in or out of hospital, at any time after randomization OR oral antibiotic therapy different from per protocol.
  Microbiological success is defined as a reduction of the pathogen found at presentation to <10^4 CFU/mL for non-catheter specimens or <10^3 for catheter specimens on urine culture.
  The EOT visit occured within 2 days of the completion of oral therapy.
Time Frame: Day 5 through Day 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Strategy 1 | Strategy 2
Number analyzed (Participants) | 24 | 27
percentage of participants | 67 [47 to 82] | 67 [49 to 82]
Statistical Analysis 1: Comparison: Strategy 1 vs Strategy 2; Test type: Other; p = 0.973, Multiple imputation using Wald method; Risk Difference (RD) = 0, 95% CI 2-sided [-26.3 to 25.3]

ADVERSE EVENTS:
Time Frame: The solicited events were collected after first dose of study product was given and until the end of therapy (EOT). If subject was on fosfomycin, solicited AEs were collected for 2 days after last dose of fosfomycin or until EOT, whichever occurred last. The unsolicited AEs were collected in participants who received at least two doses of Fosfomycin from the time of second dose of fosfomycin until the end of therapy (EOT) or 2 days after last dose of fosfomycin, whichever occurred last.
Description: Serious Adverse Events (SAEs) were only recorded in participants receiving at least two doses of fosfomycin and were not collected for other interventions. Therefore the at risk population for SAE is a subset of the safety population who received any study drug.
Groups:
- Fosfomycin: Fosfomycin was administered orally as a single 3 gram dose sachet once daily for normal kidney function or every other day for CrCl less than or equal to 20 mL/min.
- Levofloxacin: Levofloxacin was administered orally as 750 mg tablet once daily for normal kidney function, 750 mg tablet every other day for CrCl 20-49 mL/min; 500 mg tablet every other day for CrCl <20 mL/min.
- Cefixime: Cefixime was administered orally as 400mg tablet or capsule once daily for normal kidney function; 260 mg of oral suspension once daily for subjects with CrCl between 21-59 mL/min; 200 mg chewable table once daily for subjects with CrCl less than or equal to 20 mL/min.
Arm/Group | Fosfomycin | Levofloxacin | Cefixime
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/22 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/35 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 24/35 | 15/22 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosfomycin (N=35) | Levofloxacin (N=0) | Cefixime (N=0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosfomycin (N=35) | Levofloxacin (N=22) | Cefixime (N=1)
Diarrhoea (Gastrointestinal disorders) | 19 (57) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (8) | 7 (15) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (7) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (16) | 6 (14) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (10) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 7 (16) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03697993/SAP_000.pdf
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT03697993/Prot_001.pdf